CLINICAL TRIAL: NCT02134171
Title: Identification of Early Predictive Factors of Cardiac and Cerebral Involvement in Thrombotic Microangiopathies
Brief Title: Early Predictive Factors of Cardiac and Cerebral Involvement in TMA
Acronym: MATRISK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: p120118
Record Dates: First submitted 2014-03-24; First posted 2014-05-09 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Thrombotic Microangiopathies; Thrombotic Thrombocytopenic Purpura
Keywords: Thrombotic microangiopathy,; haemolytic uremic syndrome,; thrombotic thrombocytopenic purpura,; ADAMTS13,; troponin,; plasma exchange.
MeSH Terms: conditions — Thrombotic Microangiopathies; Purpura, Thrombotic Thrombocytopenic | interventions — Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Biological investigations (Experimental): From day 1 to day 3, specific blood tests will be performed (serum troponin Ic and brain natriuretic peptide [BNP]). A cardiac ultrasonography within the 4 first days and a cerebral MRI within the first 7 days after TMA diagnosis will be performed.
  Interventions: Other: Biological and imaging investigations

INTERVENTIONS:
Other: Biological and imaging investigations — From day 1 to day 3, specific blood tests will be performed (serum troponin Ic and brain natriuretic peptide [BNP]). A cardiac ultrasonography within the 4 first days and a cerebral MRI within the first 7 days after TMA diagnosis will be performed.

SUMMARY:
The aim of this study is to determine the frequency of cardiac and cerebral involvements in patients with idiopathic thrombotic microangiopathies on diagnosis. Patients will be assessed for cardiac involvement (troponin Ic level and cardiac ultrasonography) and cerebral involvement (cerebral MRI). The investigators will assess whether serum troponin Ic on diagnosis can predict morbidity and mortality of patients with a thrombotic microangiopathy at the acute phase.

The primary outcome measurement is the event free survival at day 30, as defined by death, myocardial ischemia, arrhythmia, severe cerebral injury and disease exacerbation. An increase in troponin Ic on diagnosis is defined as at least one result above 0.2 ng/ml among the three daily analyses performed after TMA diagnosis.

DETAILED DESCRIPTION:
After TMA diagnosis, patients will be treated in emergency according to standard National recommendations. Patient will be included in the study as soon as the diagnosis of TMA is performed.

From day 1 to day 3, specific blood tests will be performed (serum troponin Ic and brain natriuretic peptide [BNP]). A cardiac ultrasonography within the 4 first days and a cerebral MRI within the first 7 days after TMA diagnosis will be performed.

Our hypothesis is that an increased serum troponin Ic level on diagnosis (> 0.2 ng/ml) is a predictive feature of cardiac events or worsening at the acute phase.

At 6 months, a control cardiac ultrasonography and cerebral MRI will be performed in patients with cardiac and/or cerebral involvement on diagnosis.

122 patients are expected to be included among 30 recruiting centres in France. The total duration of inclusions is 2.5 years, and the total duration of the study is of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of thrombotic microangiopathy on the following criteria :
* A microangiopathic haemolytic anaemia (Hb< 12 g/dl, with presence of schistocytes on blood smear);
* A thrombocytopenia <150 G/l;
* No associated (precipitating) disease (HIV infection, cancer, chemotherapy, transplantation) or pregnancy;
* A written consent obtained from the patient, or from a relative for patients unable to provide the informed consent (because of cerebral involvement for example);
* Affiliation at the social insurance regimen.
* Major person

Exclusion Criteria:

* A TMA associated with an associated condition: infection with HIV (HIV) in AIDS stage, , chemotherapy, malignancy, transplantation, or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
30-day event-free survival | At 30 days
  Events include death or myocardial infarction, arrhythmia, cerebral involvement and exacerbation. Serum troponin Ic is assessed daily the 3 first days following diagnosis. Cardiac ultrasonography is performed within the 4 days following diagnosis and cerebral MRI is performed within the 7 days following the diagnosis.

SECONDARY OUTCOMES:
Cardiac trouble frequency and type at diagnosis | From day 1 to day 3 after diagnosis
Cerebral trouble frequency and type at diagnosis | From day 1 and day 7 after diagnosis
Comparison of cerebral and cardiac trouble at diagnosis between thrombotic microangiopathies type | Baseline
Description of cardiac and cerebral sequelae at M6 and reversibility frequency of diagnosis cardiac and cerebral lesions at M6 | At 6 months
Determination of cardiac and cerebral sequelae prognostic factors at M6 | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coppo, MD, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Saint Antoine, Paris, France